CLINICAL TRIAL: NCT02151552
Title: Assessing [18F](+/-)NOS Uptake With PET Imaging in Endotoxin-induced Lung Inflammation
Brief Title: Assessing NOS Uptake With PET Imaging in Lung Inflammation
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: Washington University School of Medicine (Other)
Collaborators: Doris Duke Charitable Foundation (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: DDCF 2010060-201403017
Record Dates: First submitted 2014-05-28; First posted 2014-05-30 (Estimated); Last update posted 2018-07-23 (Actual); Status verified 2018-07

CONDITIONS: Lung Inflammation
Keywords: lung inflammation; positron emission tomography; inducible nitric oxide synthase
MeSH Terms: conditions — Pneumonia | interventions — Endotoxins; Lipopolysaccharides; Fluorine-18

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Endotoxin and [18F](+/-)NOS (Experimental): All volunteers in this study will receive endotoxin in a single segment of the lung to induce mild, self-limited inflammation. They will also be imaged before and after endotoxin instillation with the novel PET tracer [18F](+/-)NOS.
  Interventions: Drug: Endotoxin (E. coli O:113, Reference Endotoxin); Drug: [18F](+/-)NOS

INTERVENTIONS:
Drug: Endotoxin (E. coli O:113, Reference Endotoxin) — The endotoxin will be reconstituted with sterile water to a final concentration of 2,000 endotoxin units/ml. The dose of 4 ng/kg will be prepared to a final volume of 2 ml and will be administered using a 5F balloon-tipped monitoring catheter inserted via a fiberoptic bronchoscope into the lateral segment of the right middle lobe of the lung on the morning of Day 2.
  Other Names: Lipopolysaccharide
Drug: [18F](+/-)NOS — 7 mCi of [18F](+/-)NOS will be injected intravenously at the start of a 60-minute dynamic PET scan acquisition

SUMMARY:
The purpose of this study is to learn more about the basic responses of the lungs to inflammation using positron emission tomography, or PET, imaging scans of the lungs. PET is a machine that detects radiation and generates pictures using a donut-shaped scanner similar in appearance to an x-ray "CAT" or computed tomography (CT) scan or an MRI. Inflammation is the way our bodies react to irritation or injury, and involves red, warm, and often painful swelling of the affected tissue. An enzyme called inducible nitric oxide synthase (iNOS) contributes to the development of lung inflammation.

DETAILED DESCRIPTION:
The investigators plan to use three radioactive tracers to produce the PET images for measuring lung inflammation: [18F](+/-)NOS (the F stands for fluorine and NOS stands for Nitric Oxide Synthase, which targets iNOS), O-15 carbon monoxide ([15O]CO), and O-15 water ([15O]H2O). The NOS tracer gives information specifically about lung inflammation, while the carbon monoxide and water tracers give information about whether the lung inflammation causes more blood or water to be retained in the area of lung inflammation.

In order to show that [18F](+/-)NOS-PET is related to the amount of inflammation, the investigators first need to create a state of controlled lung inflammation that can be measured and quantified. "Controlled lung inflammation" means a reaction in the lungs that is similar to that which occurs during lung infection (increased respiratory secretions and cough). It is "controlled" because the investigators will not be using anything alive or contagious (it does not spread from one part of the body to another, and cannot spread to another person), and a small area in only one lung will be affected. In order to created this state of controlled lung inflammation, the investigators plan to place a small amount of a purified bacterial substance called endotoxin into a single small section of the lung using a bronchoscope (a long, flexible narrow tube that is passed through the mouth into the airways of the lung). This use of endotoxin is considered investigational, and the investigators have received permission from the FDA to use endotoxin in this research study.

ELIGIBILITY:
Inclusion Criteria:

* Healthy man or woman, any race or ethnicity, age 19-44 years old
* Screening FEV1 and FVC greater than or equal to 90% of predicted
* Screening oxygen saturation by pulse oximetry greater than or equal to 97% on room air
* Capable of lying still and supine with arms raised above the head within PET/CT scanner for 2-2.5 hours
* Capable of following instructions for breathing protocol during CT portion of PET/CT scans
* Able and willing to give informed consent
* Body Mass Index (BMI) < 35

Exclusion Criteria:

* Pregnancy (confirmed by qualitative serum hCG pregnancy test)
* Lactation
* History of cardiopulmonary disease
* Currently taking any prescription medications
* History of tobacco use or illicit drug use within the past year
* Presence of implanted electronic medical device
* Enrollment in another research study of an investigational drug
* Known allergy to both trimethoprim/sulfamethoxazole and amoxicillin, Penicillin, Lidocaine, Demerol, Versed, and/or Fentanyl
* Inability to lie flat for 2-2.5 hours for PET/CT scans or follow breathing protocol instructions for the CT portion of the PET/CT
* Prior research-related radiation exposure within the past year such that participation in this study would result in exposures that exceed the limits as defined by the FDA RDRC regulations (21 CFR 361.1)

Ages: 19 Years to 44 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 3 (Actual)
Dates: Start 2014-05; Primary Completion 2018-02 (Actual); Study Completion 2018-02 (Actual)

PRIMARY OUTCOMES:
Distribution volume ratio (DVR), determined by Logan plot analysis, in the right middle lobe | Change in DVR on post-endotoxin PET scan (Day 2) from baseline (Day 1)
  Comparison of DVR by Logan plot for [18F](+/-)NOS uptake, pulmonary blood flow (PBF) and extravascular lung water (EVLW) in the regions of interest generated from scans obtained before and after endotoxin instillation and in the right and left lungs will be compared using a repeated-measures t-test, with statistical significance set at p<0.05. The DVR determined for [18F](+/-)NOS normalized for either PBF or EVLW will also be compared using a repeated-measures t-test before and after endotoxin as well as in the right and left lungs to determine whether differences in [18F](+/-)NOS uptake depend on either PBF or EVLW.

SECONDARY OUTCOMES:
Change in DVR in right middle lobe | post-endotoxin scan (Day 2) from baseline (Day 1) scan
Mean Hounsfield units (HU), measure of density on CT images, in right middle lobe and lingula | baseline PET/CT scan on Day 1 to post-endotoxin scan on Day 2
Change in HU in right middle lobe and lingula | before and after endotoxin instillation (Day 1 to Day 2)
Bronchoalveolar lavage (BAL) cell counts (including total nucleated and neutrophil counts) | 6 hours post-endotoxin instillation
Number and percent of iNOS-stained BAL cells by flow cytometry | 6 hours post-endotoxin instillation
Number and percent of 3-nitrotyrosine-stained cells on biopsy | 6 hours post-endotoxin instillation
Change in exhaled nitric oxide (ENO) levels | before and after endotoxin instillation (Day 1 to Day 2)
Regional PBF and EVLW in right middle lobe and lingula | before and after endotoxin (Day 1 to Day 2)
Number of iNOS positive cells from brushing cytospins | 6 hours post-endotoxin instillation

CONTACTS AND LOCATIONS:
Overall Officials: Delphine Chen, MD, Principal Investigator — Washington University School of Medicine
Locations (1):
- Washington University School of Medicine / Barnes-Jewish Hospital, St Louis, Missouri, United States